CLINICAL TRIAL: NCT07241598
Title: Cognitive-motor Training in Community-dwelling Older People With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Neuroscience Research Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-CIRB 2025/147.0205
Record Dates: First submitted 2025-05-31; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: mild cognitive impairment; MCI; dementia; cognitive training; older adults; older people; community-dwelling; cognitive-motor training; RCTs; exergaming program; A randomised controlled trial; falls; falling; preventing falls; risk of falls
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: This research will use a single-blind randomized controlled trial (RCT) to assess the effects of the Smart±step cognitive-motor training program compared to usual care. The study will recruit community-dwelling older adults with MCI, defined using Petersen's criteria and objective cognitive measures such as the Montreal Cognitive Assessment (MoCA). Participants will be randomly allocated to either the Smart±step intervention group or the control group, with the intervention group receiving 120 minutes of Smart±step training per week for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group will receive Smart±step cognitive-motor training for 12 weeks (Experimental): Participants allocated to the intervention group will be provided with the Smart±step system and recommended to exercise at least 120 minutes per week for 12 weeks.
  Interventions: Device: Smart±step cognitive-motor training
- The control group (No Intervention): The control group will receive usual care and existing healthy living information.

INTERVENTIONS:
Device: Smart±step cognitive-motor training — 12 weeks of Smart±step cognitive-motor training for older people with mild cognitive impairment (MCI)
  Arms: The intervention group will receive Smart±step cognitive-motor training for 12 weeks

SUMMARY:
As the global population ages, the prevalence of mild cognitive impairment (MCI) among older adults, which ranges from 5% to 40%, is expected to rise. MCI significantly increases the risk of developing Alzheimer's disease and is associated with a heightened risk of falls, with evidence suggesting that individuals with MCI have a fall risk five times greater than their cognitively intact peers. While cognitive and physical impairments in MCI are recognized, targeted interventions addressing both aspects are needed.

This study aims to evaluate the effectiveness of the Smart±step exergaming program, an interactive system combining cognitive and motor training through computer-based stepping tasks, in reducing risk of falls, fall rate and improving physical, cognitive, psychological, neurophysiological, and quality of life outcomes in community-dwelling older adults with MCI. Previous research indicates that combined cognitive-motor interventions can improve balance and cognitive outcomes, but evidence on their efficacy in reducing falls is limited.

The study will assess whether the Smart±step program, previously shown to be effective in cognitively healthy populations, can also significantly reduce risk of fall, fall rates and enhance overall function in older people with MCI. If successful, the program could offer substantial benefits by lowering fall-related costs and disabilities, with potential for global adaptation and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Older people with MCI will be identified based on the core criteria outlined by the diagnostic scheme of MCI by Petersen and the National Institute on Aging-Alzheimer's Association and as follows: Subjective cognitive complaints (SCCs) will be assessed using four commonly endorsed items from Slavin et al., with a total score ≥3 indicating SCCs. Objective cognitive impairment will be determined using the Thai version of the Montreal Cognitive Assessment (MoCA), with inclusion criteria defined as MoCA scores of 20-25 for individuals with ≤12 years of education and 21-25 for those with >12 years. Functional ability will be evaluated using the Bayer Activities of Daily Living Scale (B-ADL), with scores <3 indicating no impairment. Participants with MoCA scores <20 (≤12 years education) or <21 (>12 years) will be excluded to rule out dementia. Individuals meeting all four criteria-subjective complaints, objective cognitive impairment, preserved functional abilities, and absence of dementia-will be classified as having MCI.
* Aged 60 years or more.
* Thai-speaking language and able to read or understand the Thai language
* Able to walk 10m independently (without a walking aid)

Exclusion Criteria:

* Having had a stroke in the last 2 years.
* Having a progressive neurodegenerative disorder e.g. Parkinson's disease, Multiple sclerosis, amyotrophic lateral sclerosis (ALS).
* Individuals who are blind, deaf, or amputees, whether the condition is congenital or acquired.
* A medical condition that would interfere with the safety and conduct of the training and testing protocol or interpretation of the results, such as:

  1. Musculoskeletal conditions e.g. severe pain of lower extremities (pain score > 4/10), recent TKR/THR (less than or equal to 12 months after operation) and recent fracture (12-months).
  2. Cardiopulmonary conditions e.g. unstable angina, uncontrolled hypertension.
  3. Metabolic conditions e.g. severe or poorly controlled diabetes.
  4. Mental health conditions e.g. severe or poorly controlled depression or psychiatric condition.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Stroop stepping test | Baseline, 3-month reassessment, 6-month post-intervention , and 12-month post-intervention
  Stroop stepping test (SST) will be used to measure the ability to perform accurate stepping with response inhibition using the Choice Stepping Reaction Time Test. This equipment consists of a custom-made dance pad (150×90cm) which is connected to a computer and display screen (1280 × 768 pixels; 60 Hz; 58 cm). The test will start when an arrow shows in the centre of the monitor pointing in one of four directions (up, down, left and right) that matched the four possible step directions (forward, backward, left and right). A word indicating a different direction will be written inside the arrow. Participants will be instructed to 'Step by the word' and will have to inhibit the response indicated by the arrow's orientation. Four practice trials are not included in the score and 20 trials will be administered randomly by the directions of word and orientation. The average time (ms) and number of errors will be recorded.
Physiological profile assessment | Baseline, 3-month reassessment, 6-month post-intervention , and 12-month post-intervention
  Fall risk will be assessed with the Physiological Profile Assessment (PPA), which provides a total fall-risk score from five measures: edge contrast sensitivity, lower limb proprioception, lower limb strength, simple hand reaction time, and postural sway. Edge contrast will be tested with the Melbourne Edge Test, proprioception by toe alignment with eyes closed, strength by maximal leg extension against a spring gauge, reaction time by response to a light stimulus via modified mouse, and sway by swaymeter during 30-second standing trials on firm and foam surfaces with eyes open and closed. PPA assessments will be used to calculate the PPA fall-risk score, with higher scores indicating poorer physical performance and greater risk of falling.

SECONDARY OUTCOMES:
Timed Up and Go Test | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Mobility will be measured using the Timed Up and Go Test (TUG). Participants will be instructed to rise from a standard chair with arms, walk a distance of three metres at usual pace, turn around, walk back to towards the chair, and sit down again. The time in seconds will be recorded beginning at the instruction "go" and stopping when the participant is seated. One practice trial is not included in the score and therefore the mean of 2 trials will be calculated and used for statistical analysis. Dual task test will be assessed using TUG test combined with a verbal fluency task by naming animals. Participants will be instructed to rise from a standard chair with arms, walk a distance of three metres, turn around, walk back to towards the chair, and sit down again. In the meantime, participants will have to name as many animals as they can. The time to complete the TUG will be recorded in seconds. The mean of 2 trials will be calculated and used for statistical analysis.
Short Physical Performance Battery | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Lower extremity functioning will be assessed using the Short Physical Performance Battery (SPPB). The scores range from 0 to 12 (higher score indicating better performance) and are based on performance on three tasks including gait speed, chair stand, and static standing balance with different three standing positions.
30s-Chair-Stand Test | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  The 30-second Chair Stand Test will be used to assess lower body strength and endurance, particularly of the hip and thigh muscles important for daily mobility and fall prevention. Using a standard armless chair about 43-45 cm high, participants will sit with feet flat and arms crossed over the chest. At the signal "go," they will repeatedly stand to full extension and sit back down as many times as possible within 30 seconds without using their arms. The score will be the total number of full stands completed before time expires; partial rises will not be counted. Higher counts will indicate greater lower limb strength and functional capacity.
Trail-Making Test (TMT) Part A and B and the Controlled Oral Word Association Test (COWAT) | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Executive function will be assessed using Trail-Making Test (TMT) Part B and the Controlled Oral Word Association test (COWAT). For TMT Part B, participants will be instructed to draw a line to connect consecutive numbers in numerical order and letters in alphabetical order in an alternating sequence (e.g., 1-ก-2-ข-3-ค) as quickly and correctly as possible. For the COWAT, participants will have to generate as many words as possible in a 60s timeframe starting with F, then A, then S. The score will be calculated by the number of words correctly iterated. Attention and processing speed will be assessed using Trail-Making Test (TMT) Part A and the digit symbol Substitution. For TMT Part A, participants will be instructed to draw a line to connect consecutive numbers in numerical order as quickly and correctly as possible (e.g., 1-2-3).
Semantic fluency | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Semantic fluency will be assessed using the animals naming test. Participants will be asked to generate as many animals as they can within 60 second. The total score will be calculated from the maximum number of animals listed.
The modified switching verbal fluency test | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  The modified switching verbal fluency test (mSVF) will be a cognitive flexibility test. In this test, participants will be required to alternately present words from two categories, fruits and animals, as many as possible within a 1-minute period. The researcher will record the correct word count for each category.
The digit symbol substitution | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  For the digit symbol substitution, participants will be instructed to match symbols to numbers according to a key located on the top of the paper test. Participants will have to copy the symbol into spaces below a row of numbers. The score will be calculated by the total number of correct symbols within the allowed time, usually 90 to 120 seconds.
The Digit Span test | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Short-term auditory memory and working memory will be measured using the two parts of the Digit Span test: Digits Forward and Digits Backward. These will be administered separately. The digits will be presented at a rate of one per second. In Digits Forward (DSF), the patient is required to repeat the digits in the same order as presented. In Digits Backward (DSB), the patient is required to repeat the digits in reverse order. Participants will listen to a series of numbers presented at 1 number per second and repeat them either in the same order (DSF) or in reverse (DSB). For example, after hearing "6, 9, 4, 7," participants will repeat "6, 9, 4, 7" (DSF) or "7, 4, 9, 6" (DSB). Numeric sets will range from 2 to 10 digits. Each set will be tested three times. If participants correctly recall the sequence at least twice, they will pass that set. Failure to do so will result in stopping the test.
Short Falls Efficacy Scale international | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Fear of falling will be assessed using short Falls Efficacy Scale international (Short FES-I). The Short FES-I version which is an interview-based questionnaire contains 7 activities of daily living. The level of concern about falling through a combination of pictures and matching short phrases is scored on a 4-point scale (1 = not at all concerned to 4 = very concerned). The total score ranges from 7 to 28.
Thai Geriatric Depression Scale | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Symptoms of depression will be assessed using Thai Geriatric Depression Scale (TGDS). The short form of TGDS is a 15-item self-report questionnaire that inquiries about depressive emotion in daily situations experienced in the past week. Participants will rate each item as yes or no, scores range from 0 to 15, with higher scores indicating greater symptom severity.
Thai Geriatric Anxiety Scale | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Anxiety symptoms will be assessed using Goldberg Anxiety Scale (GAS). The GAS consists of 9-item for self-rating of anxiety experienced in the past month which includes affective and somatic symptoms of anxiety. The score will be rated as yes (1) or no (0) answers with a total score ranging from 0 to 9 which higher scores substantially increase the probability of a significant anxiety disorder.
Electroencephalogram (EEG) | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Participants will perform electroencephalogram (EEG) recordings during resting-state. In the resting-state, each participant will seat in a comfortable chair in a relaxed position during the EEG measurement, which consists of 5-minute session for eyes opened and eyes closed conditions. The EEG signals will be recorded during resting state using an eegoTMmylab ANT Neuro (32-electrodes EEG cap). The EEG recording will use a sampling rate of 512 Hz and a notch filter of 50 Hz. A software filter will set to bandpass with a low pass of 0.3 Hz and a high pass of 100 Hz. The impedance of the electrode-skin interface will keep below 20kΩ, as recommended in prior scholarship. The EEG instrument consisted of 32 channels at the recording of position includes Fp1, Fpz, Fp2, F7, F3, Fz, F4, F8, FC5, FC1, FC2, FC6, T7, T8, C3, Cz, C4, CP5, CP1, CP2,CP6, P3, P7, Pz, P4, P8, POz, O1, Oz, O2, M1, M2, CPz (reference electrode), and AFz (ground electrode).
Event Related Potential (ERP) | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Participants will perform the event-related potentials (ERPs) recordings during Go/No-go task (using 4 images) in response to visual stimuli. Participants will have the brain activity measured with an electroencephalography (EEG) cap while performing an image-viewing task. The cap will record the brain signals as participants view images and respond by pressing a pedal with their's dominant foot. Participants will complete practice pedal presses to become familiar with the response before the actual test. When participants see image "(1)" or "(3)" they should press the pedal; when they see image "(2)" or "(4)" they should not press the pedal. The picture stimuli will present in random order during each trial, and each trial lasted 2-minutes. Participants will give a 5-minute rest between trials, and the duration of the two experiments was 40 minutes.
Physical Activity Scale for Elderly Thai version | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  The Physical Activity Scale for the Elderly (PASE) Thai-version evaluates physical activity through 10 questions covering walking, exercise, household chores, and work. Participants will report activity type, frequency, and duration over the past week. Scores are calculated by multiplying activity frequency and duration by assigned weights. Activities like chores and work are scored based on average daily hours, adjusted by weights; sedentary tasks score 0. The total score, ranging from 0 to 400, excludes sitting activities.
WHOQOL-BREF-THAI | Baseline, 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  The participants' QOL will also be evaluated by using the WHOQOL-BREF-Thai questionnaire that can be assessed by self-report. In situations that the participants cannot read, the assessor will read for them, and they will have to choose the answer by themselves. The WHOQOL-BREF questionnaire has two types of questions: perceived objective and self-report subjective, and it includes four components of well-being: physical, psychological, social, and environmental. Each item is scored from 1-5. This Thai version has a good internal consistency with Cronbach's alpha 0.84. The higher score indicates better QOL.
Falls rate (12 month prospective falling record) | 3-month reassessment, 6-month post-intervention, and 12-month post-intervention
  Each participant will be given weekly fall diaries to mark any falls during the study period. A fall is defined as "an unexpected event in which the person comes to rest on the ground, floor, or lower level". If fall data is not received, telephone calls will be used to obtain fall data.
System Usability Scale (intervention group only) | Baseline and 3-month reassessment
  At the completion of the Smart±step training (3 months and 6-months), participants will rate the usability of the Smart±step training using the System Usability Scale (SUS): SUS scores of 50-70 are acceptable, 71-85 are good to excellent, >85 are excellent usability, and <50 are considered unacceptable.
Physical Activity Enjoyment Scale (PACES) Thai version | Baseline and 3-month reassessment
  Enjoyment during engaging in the Smart±Step training exercise will assess using Physical Activity Enjoyment Scale (PACES) Enjoyment Scale (PACES). The PACES is an 8-item scale questionnaire that measures the level of enjoyment using a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scores for enjoyment were obtained through the sum of PACES scores. A higher score indicates a greater level of enjoyment.
Sessions and time recorded by training system and logbook record | Baseline and 3-month reassessment
  All participants will be instructed to complete a logbook immediately after each exercise session to ensure data accuracy. Adherence to the intervention will be calculated as the percentage of Smart±Step sessions attended, using the formula: ((n/24 sessions) x 100). Any adverse events occurring during the study, such as injuries, falls, fatigue, or other exercise-related issues, will be documented. Furthermore, participants will be asked about their training experiences and any health issues at every follow-up point throughout the study. They will also be encouraged to contact the research team at any time with questions or concerns.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-11-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT07241598/Prot_SAP_ICF_000.pdf